CLINICAL TRIAL: NCT07327138
Title: A Multi-center, Assessor-blinded, Randomized, Parallel Group, Superiority Trial Evaluating the Efficacy of Home-based Laughter and Fun Yoga as an Adjunct for Pain Reduction in Pediatric Oncology Patients Receiving Chemotherapy.
Brief Title: Children's Laughter and Fun Yoga as Adjunctive Pain Relief Following Chemotherapy.
Acronym: CLAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahaa Bou Dargham (Other)
Collaborators: Beirut Arab University (Other); Hammoud Hospital University Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Bahaa Bou Dargham, Lecturer of Anesthesia, Beirut Arab University
Organization: Beirut Arab University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-Jun2025-IX
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia ALL
Keywords: Acute Lymphoblastic Leukemia; Chemotherapy; Steroids; Pediatric Oncology; Pain Management; Cancer-related Pain; Laughter Therapy; Yoga Therapy; Non-pharmacological Intervention; Home-based Intervention; Supportive Cancer Care
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Agnosia; Cancer Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter and Fun Yoga Plus Usual Care (Experimental): Participants randomized to this arm will receive the Magic Box Laughter and Fun Yoga Program in addition to usual care. The intervention is a structured, home-based program delivered over six consecutive days and supported by guided videos and daily activity packages. On the hospital visit day, parents receive an introduction video, the Magic Box, and six numbered packages, along with instructions and daily follow-up arrangements. Each day, parents receive a short video guiding age-appropriate activities that combine gentle fun yoga, breathing exercises, laughter-based exercises, and playful activities using materials provided in the daily packages. Parents actively supervise and participate with the child throughout the program. The intervention concludes with a celebratory session focused on positive affirmation and engagement. All participants continue to receive standard medical and supportive pain management according to institutional protocols.
  Interventions: Behavioral: Laughter and Fun Yoga Program
- Usual Care Only (No Intervention): Participants randomized to this arm will receive usual care only, consisting of routine pharmacological and supportive pain management according to each participating center's pediatric oncology protocols. This may include analgesic medications, such as opioids if clinically indicated, as well as general supportive measures including rest, hydration, and comfort care. No structured laughter therapy, yoga activities, or other psychosocial interventions will be provided as part of the study. All participants in this arm will continue to receive standard medical care throughout the study period.

INTERVENTIONS:
Behavioral: Laughter and Fun Yoga Program — This intervention consists of a structured, home-based laughter and fun yoga program delivered over six consecutive days. The program combines guided video-based sessions with daily activity packages containing materials for age-appropriate playful activities. The activities include gentle fun yoga movements, breathing exercises, laughter-based exercises, guided play, and positive affirmation. Parents or caregivers supervise and actively participate with the child throughout the program. The intervention is designed to be non-invasive, low intensity, and safe for children receiving chemotherapy, and it is provided in addition to standard medical and supportive care.
  Arms: Laughter and Fun Yoga Plus Usual Care

SUMMARY:
The goal of this clinical trial is to learn if a home-based program that combines laughter and fun yoga can help lower pain in children receiving chemotherapy. The study focuses on children with acute lymphoblastic leukemia who experience pain during treatment with chemotherapy and steroids.

The main questions this study aims to answer are:

1. Does adding laughter and fun yoga to usual care lower pain levels in children receiving chemotherapy?
2. Does this program reduce the need for strong pain medicines, such as opioids?
3. Does the program help improve mood, anxiety, and sleep during treatment?

Researchers will compare children who receive laughter and fun yoga plus usual care with children who receive usual care alone to see if the program works.

Participants will:

1. Be randomly assigned to either the laughter and fun yoga group or the usual care group
2. Take part in the study during a 6-day period after receiving their chemotherapy treatment
3. Have their pain measured once each day using a child-friendly pain scale
4. Have parents answer short questions about pain medicine use, mood, anxiety, and sleep

The laughter and fun yoga activities are gentle, safe, and designed to be done at home with the help of a parent. All participants will continue to receive their regular medical care throughout the study.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, parallel-group clinical trial evaluating the effectiveness of a structured home-based laughter and fun yoga intervention as an adjunct to standard care for the management of chemotherapy-related pain in children with acute lymphoblastic leukemia.

Participants are enrolled during routine chemotherapy visits and undergo baseline assessment prior to randomization. Using a 1:1 allocation ratio, participants are assigned to either the intervention group or the control group. Randomization is performed to ensure balanced group allocation across participating study centers.

The intervention consists of a structured program delivered at home over a six-day period. It integrates gentle, age-appropriate yoga movements, breathing exercises, laughter-based activities, and guided play. The activities are designed to be non-invasive, low intensity, and safe for children undergoing chemotherapy. Parents or caregivers supervise and actively participate in the sessions to support engagement and ensure safety. The intervention is intended to complement, not replace, standard medical care.

Participants assigned to the control group receive standard care only, which includes routine pharmacological and supportive pain management according to institutional protocols at each participating center. No structured laughter or yoga activities are provided to the control group during the study period.

Outcome data are collected through brief daily assessments conducted during the intervention period. Pain is assessed daily using a validated, child-friendly pain rating scale. Additional information on pain medication use and selected psychosocial outcomes is collected through parent-reported measures. Data collection procedures are designed to minimize participant burden and integrate smoothly into routine care.

The primary objective of the study is to determine whether the addition of a structured, non-pharmacological home-based intervention can lower pain intensity during chemotherapy. Secondary objectives include evaluating the potential impact of the intervention on pain medication use and overall well-being. The findings of this study may help inform supportive care strategies for children undergoing cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-10 years.
* Medically diagnosed with acute lymphoblastic leukemia (ALL) and currently receiving chemotherapy that includes dexamethasone pulses during the maintenance phase.
* Clinically stable and able to participate in gentle, low-intensity yoga movements as determined by the treating physician.
* At least one parent or legal guardian willing and able to supervise and participate in the home-based intervention sessions.
* Written informed consent from parent/legal guardian, with age-appropriate assent from the child.

Exclusion Criteria:

* Recent major surgery (within the past 2 weeks) that may limit safe participation in gentle activity.
* Severe uncontrolled medical conditions (unstable vital signs, decompensated cardiac or respiratory disease, uncontrolled epilepsy) that may place the child at risk during light movement or laughter.
* Severe visual, hearing, or cognitive impairment preventing engagement with video-based instructions and exercises.
* Physical limitations or musculoskeletal injuries that prevent participation in the intervention.
* Any other condition that, in the judgment of the treating physician, would interfere with safe participation or adherence.
* Currently enrolled in another interventional clinical trial for pain management.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Pain Intensity on Days 5 and 6 | Days 5 and 6 post chemotherapy and steroid administration
  Pain intensity will be assessed using the Wong-Baker FACES Pain Rating Scale (FPS-R), a validated, child-friendly self-report tool that uses facial expressions anchored to numerical values from 0 (no pain) to 10 (worst pain). Pain will be assessed once daily at a consistent time using a standardized parent-read script, and the child will select the face that best represents their pain at that moment. Scores will be recorded immediately after assessment. The primary endpoint is defined as the average pain score measured on Day 5 and Day 6 post chemotherapy and steroid administration, corresponding to the expected peak dexamethasone-related pain window. If only one of these two measurements is available, that value will be used as the primary outcome.

SECONDARY OUTCOMES:
Daily pain trajectory (Wong-Baker FACES) | From Day 0 to Day 6 post chemotherapy and steroid administration
  Daily pain will be measured using the Wong-Baker FACES Pain Rating Scale (0, 2, 4, 6, 8, 10) at a fixed evening window (17:00-20:00) on Days 0-6 to characterize the day-by-day trajectory of pain during the dexamethasone period. At each assessment, a standardized script will be read by the parent under researcher guidance, and the child will select the face that best represents their pain "right now." If no clear response is given, the script may be repeated once without prompting toward any choice. Scores will be recorded immediately on the CRF with date and time. This outcome provides a daily series of FPS-R values across the 7-day observation window, enabling description of within-week pain patterns and comparison of peak timing and magnitude between groups, complementary to the primary endpoint (Day 5-6 average).
Analgesic use (opioids only) | From Day 0 to Day 6 post chemotherapy and steroid administration
  Opioid analgesic use will be assessed during the dexamethasone and chemotherapy period, as non-opioid analgesics are not routinely used during this phase. Opioid exposure will be measured by converting all administered opioid doses to oral morphine milligram equivalents (MME), including cumulative 6-day MME and weight-adjusted MME per kilogram. Additional measures include time from chemotherapy and dexamethasone administration to first rescue opioid dose, number of rescue opioid doses, and the proportion of participants requiring any opioid analgesia. Emergency department visits for pain control during the study period will also be recorded, including opioid administration and disposition when applicable.
Depression | Day 0 and Day 6
  Depressive symptoms will be assessed using the Arabic Short Mood and Feelings Questionnaire - Parent version (SMFQ-P), a 13-item parent-reported questionnaire that evaluates core depressive symptoms such as sadness, loss of interest, irritability, fatigue, guilt, and low self-esteem. Each item is rated on a 3-point scale ("not true," "sometimes true," "true"), with total scores ranging from 0 to 26; higher scores indicate greater depressive symptom severity. The Arabic SMFQ-P has been validated in Lebanon and is appropriate for use in research settings. The questionnaire will be administered to parents at baseline (Day 0) and at the end of the intervention period (Day 6). For younger children, the tool will be completed as a parent-proxy measure focusing on observable mood and behavior.
Anxiety | Day 0 and Day 6
  The SCARED-5 (5-item Screen for Child Anxiety Related Emotional Disorders) is a brief parent-report screening tool used for youth anxiety. Although an Arabic validation of the short version is not yet available, the full Arabic SCARED-P (41-item parent version) has demonstrated excellent psychometric properties in Lebanon (a = 0.92, convergent validity with SDQ Emotional, discriminant validity). The SCARED-5 has undergone a recent psychometric evaluation, showing strong internal consistency, single-factor structure, good correlation with the full scale, and a suggested cutoff score of ≥ 2 for identifying anxiety. Based on this evidence, we will use the Arabic version of the items from the validated full SCARED-P, structured as the SCARED-5, and apply a clinical alert threshold of ≥ 2. In younger children (age <6), scores will be treated as exploratory and interpreted with caution.
Sleep Quality | Day 0 and Day 6
  Sleep will be assessed using the Arabic Sleep Disturbance Scale for Children (SDSC), a 26-item parent-reported questionnaire that evaluates common pediatric sleep problems, including difficulties with sleep initiation and maintenance, breathing-related sleep disturbances, arousal disorders, excessive daytime sleepiness, and sleep-wake transition problems. Each item is rated on a 5-point scale, with higher total scores indicating greater sleep disturbance. The SDSC will be administered at baseline (Day 0) and at the end of the intervention period (Day 6). The primary sleep outcome is the change in total SDSC score from baseline to Day 6. For younger children, results will be exploratory. Participants with markedly elevated scores will be flagged and referred to the treating physician for clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa W Bou Dargham, MD, Principal Investigator — Beirut Arab University and Hammoud Hospital University Medical Center
Locations (1):
- Hammoud Hospital University Medical Center, Sidon, Lebanon

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. This study involves pediatric participants and includes sensitive clinical and psychosocial information. Data sharing is not planned due to privacy considerations and local institutional and ethical requirements.